CLINICAL TRIAL: NCT00101153
Title: A Phase I Study Of Therapy With The Farnesyl Transferase Inhibitor R115777 (Zarnestra) Combined With Conventional Induction And Consolidation Chemotherapy For Previously Untreated Patients Over Age 55 With Acute Myeloid Leukemia (AML)
Brief Title: Tipifarnib, Cytarabine, and Daunorubicin in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PMH-PHL-026; CDR0000405840 (Registry Identifier: PDQ (Physician Data Query)); NCI-6670
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Leukemia
Keywords: adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Daunorubicin; tipifarnib

ARMS (1):
- Tipifarnib with conventional induction and consolidation (Experimental)
  Interventions: Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: tipifarnib

INTERVENTIONS:
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: tipifarnib

SUMMARY:
RATIONALE: Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cytarabine and daunorubicin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving tipifarnib together with cytarabine and daunorubicin may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of tipifarnib when given with cytarabine and daunorubicin in treating older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of tipifarnib when administered with cytarabine and daunorubicin in older patients with previously untreated acute myeloid leukemia.
* Determine the toxicity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of tipifarnib.

Induction therapy (1 course): Patients receive cytarabine IV continuously on days 1-7, daunorubicin IV on days 6-8, and oral tipifarnib twice daily on days 6-15 in the absence of unacceptable toxicity. Patients achieving complete remission proceed to consolidation therapy.

Consolidation therapy (1 course): After hematologic recovery, patients begin consolidation therapy 35-60 days after the start of induction therapy. Patients receive cytarabine, daunorubicin, and tipifarnib as in induction therapy.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A total of 10 patients are treated at the recommended phase II dose.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 3-28 patients will be accrued for this study within 1.5-22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)

  * All subtypes, except acute promyelocytic leukemia, are allowed
  * At least 20% bone marrow or peripheral blood blasts OR biopsy-confirmed extramedullary disease
* No cerebrospinal fluid involvement

PATIENT CHARACTERISTICS:

Age

* 56 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* See Disease Characteristics
* WBC < 100,000/mm^3 (treatment with hydroxyurea allowed)

Hepatic

* Bilirubin ≤ 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 2.0 times ULN

Renal

* Creatinine < 1.7 mg/dL OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* LVEF ≥ 50%
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Immunologic

* HIV negative
* No history of allergic reaction attributed to compounds of similar chemical or biologic composition to tipifarnib or imidazole drugs (e.g., ketoconazole, clotrimazole, or miconazole)
* No ongoing or active infection

Other

* Not pregnant
* Fertile patients must use effective contraception
* Able to swallow oral medications
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for AML except hydroxyurea for cytoreduction
* More than 4 weeks since prior chemotherapy except hydroxyurea (6 weeks for nitrosoureas or mitomycin) and recovered

  * At least 24 hours since prior hydroxyurea

Endocrine therapy

* No concurrent dexamethasone

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy > 3,000 cGy to marrow-producing areas

Surgery

* Not specified

Other

* No other concurrent investigational agents
* No other concurrent antileukemic agents
* No concurrent treatment with any of the following:

  * Ketoconazole
  * Itraconazole
  * Voriconazole
  * Clarithromycin
  * Erythromycin
  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Cyclosporine
  * Pimozide
  * Warfarin
  * Grapefruit juice
  * Simvastatin
  * Lovastatin
  * Atorvastatin
* No concurrent magnesium- or aluminum-containing antacids within 2 hours before or after tipifarnib administration

Min Age: 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-04; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of tipifarnib when administered with cytarabine and daunorubicin | minimum of 30 days per treatment cycle
Toxicity | All cycles
Pharmacokinetics | Day 6

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Brandwein, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario

REFERENCES:
- [Result] Brandwein JM, Leber BF, Howson-Jan K, Schimmer AD, Schuh AC, Gupta V, Yee KW, Wright J, Moore M, MacAlpine K, Minden MD; NCI CTEP Protocol 6670. A phase I study of tipifarnib combined with conventional induction and consolidation therapy for previously untreated patients with acute myeloid leukemia aged 60 years and over. Leukemia. 2009 Apr;23(4):631-4. doi: 10.1038/leu.2008.341. Epub 2008 Dec 18. PMID 19092853